CLINICAL TRIAL: NCT03142503
Title: Effectiveness of a Dietary Intervention Program on Disease Activity, Metabolism and Oxidative Stress in Patients With Psoriatic Arthritis and Psoriasis Activity: A Clinical, Randomized, Placebo-controlled Trial
Brief Title: The DIET Trial - Dietetic Intervention in Psoriatic Arthritis
Acronym: DIET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Marcelo M Pinheiro, Assistant Professor, Federal University of São Paulo
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2012/18701-2
Record Dates: First submitted 2017-04-06; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Arthritis, Psoriatic; Metabolic Syndrome
Keywords: psoriatic arthritis; psoriasis; body composition; DXA measurements; spondyloarthritis; diet therapy; adipose tissue
MeSH Terms: conditions — Arthritis, Psoriatic; Metabolic Syndrome; Psoriasis; Spondylarthritis | interventions — Diet; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator): Soybean supplementation
  Interventions: Dietary Supplement: Placebo
- Diet + placebo (Active Comparator): Soybean supplementation and diet intervention
  Interventions: Dietary Supplement: Diet + placebo
- Diet + Supplementation (Experimental): Omega 3 and diet intervention
  Interventions: Dietary Supplement: Diet + supplementation

INTERVENTIONS:
Dietary Supplement: Diet + supplementation — Supplementation of 1g of fish oil, 3 time a day, and hypocaloric diet (-500 calories) for 12 weeks, to evaluate weight loss, antioxidant markers and disease activity.
  Arms: Diet + Supplementation
Dietary Supplement: Diet + placebo — Supplementation of 1g of soybean oil, 3 times a day, and hypocaloric diet (-500 calories) for 12 weeks, to evaluate weight loss, antioxidant markers and disease activity.
  Arms: Diet + placebo
Dietary Supplement: Placebo — Supplementation of 1g soybean oil, 3 times a day.
  Arms: Placebo

SUMMARY:
Psoriasis (Ps) and psoriatic arthritis (PsA) are associated with increased risk of metabolic syndrome (MetS), body fatness and cardiovascular risk. Additionally, oxidative stress and inflammation are also contributing mechanisms on Ps and PsA. However, little is known about the influence of diet and micronutrients on the main outcomes of these diseases. The aim of the investigators is to evaluate the effectiveness of an intervention diet program on disease activity, metabolic profile and oxidative stress inpatients with Psoriasis and Psoriatic Arthritis.

ELIGIBILITY:
Inclusion Criteria:

* patients with psoriatic arthritis, according to the Classification Criteria of Psoriatic Arthritis (CASPAR)

Exclusion Criteria:

* lack of written informed consent;
* age < 18 years old;
* history of gastrointestinal, endocrine, pulmonary, kidney, hepatic, and neuromuscular diseases, as well as HIV-positive;
* pregnant or breast-feeding women;
* previous history of cancer;
* use of steroids, protein supplements, vitamins, multivitamins, or antioxidants.
* Specific medications to PsA and physical activity were required to be stable for the last 3 months to be included in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2013-01-21 (Actual); Primary Completion 2015-03-16 (Actual); Study Completion 2015-06-22 (Actual)

PRIMARY OUTCOMES:
Disease activity | 12 weeks
  To evaluate the increase of Minimal Disease Activity (MDA) after intervention

SECONDARY OUTCOMES:
Fat Mass | 12 weeks
  To analyze the decrease of Fat Mass Index (kg/m^2)
Lean Mass | 12 weeks
  To evaluate the increase of Muscle Mass (kg)
Waist circumference | 12 weeks
  To observe the improvement of waist circumference (cm)
Body Mass Index | 12 weeks
  To analyze the improvement of Body Mass Index (kg/m^2)
Glycation markers | 12 weeks
  To analyze the decrease of receptor for advanced glycation end products receptor (RAGE)
Anti-inflammatory marker | 12 weeks
  To analyze the increase of adiponectin
Lipidic Peroxidation | 12 weeks
  To analyze the improvement of malondialdehyde (TBARs)
Inflammatory markers | 12 weeks
  To observe the improvement of LDL fractions
Cutaneous activity | 12 weeks
  To evaluated the reduction in cutaneous activity, evaluated by PASI (Psoriasis Area Severity Index)
Articular activity | 12 weeks
  To evaluate the decrease of articular activity, evaluated by DAS28-CRP (Disease Activity Score-C reactive protein) and DAS28-ESR (Disease Activity Score-Erythrocyte Sedimentation Rate).

REFERENCES:
- [Derived] Scherer D, Leite BF, Morimoto MA, Oliveira TL, Klemz BNC, Freitas RAMS, Pappiani C, Damasceno NRT, Pinheiro MM. Nutritional effect on lipoproteins and their subfractions in patients with Psoriatic Arthritis: a 12-week randomized trial-the DIETA trial. Adv Rheumatol. 2024 Jun 13;64(1):47. doi: 10.1186/s42358-024-00389-5. PMID 38872193
- [Derived] Leite BF, Morimoto MA, Gomes CMF, Klemz BNC, Genaro PS, Shivappa N, Hebert JR, Damasceno NRT, Pinheiro MM. Dietetic intervention in psoriatic arthritis: the DIETA trial. Adv Rheumatol. 2022 Apr 6;62(1):12. doi: 10.1186/s42358-022-00243-6. PMID 35387686